CLINICAL TRIAL: NCT01974661
Title: A Phase I Open-label Study to Evaluate Safety and Immunologic Response of COMBIG-DC Administered Intra-tumorally in Patients With Hepatocellular Carcinoma
Brief Title: Phase I Safety Study of Dendritic Cell Vaccine to Treat Patients With Hepatocellular Carcinoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mendus (Industry)
Collaborators: Uppsala University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IM-102; 2013-001787-31 (EudraCT Number)
Record Dates: First submitted 2013-10-21; First posted 2013-11-01 (Estimated); Last update posted 2017-09-29 (Actual); Status verified 2017-09

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- COMBIG-DC (Experimental): COMBIG-DC (allogeneic dendritic cells) Cancer Vaccine 3 vaccinations: 5, 10 or 20 million cells per injection
  Interventions: Biological: COMBIG-DC (ilixadencel)

INTERVENTIONS:
Biological: COMBIG-DC (ilixadencel) — Allogenic dendrite-cell based therapeutic vaccine
  Other Names: ilixadencel

SUMMARY:
The primary objective of this study is to answer the question "Is it possible to inject the COMBIG-DC vaccine in a hepatic tumor without getting unacceptable side effects"?

DETAILED DESCRIPTION:
Patients diagnosed with hepatocellular carcinoma will get COMBIG-DC vaccinations at three occasions with 2-3 weeks and 3-5 weeks between vaccination 2 and 3 respectively. Adverse events will be registered until 6 months after last vaccination, as well as changes in vital signs (heart rate, blood pressure and body temperature) and lab parameters. Immunologic response will be evaluated by measuring immunologic markers in blood. The size of the tumor/tumors will be evaluated after 3 and 6 months and thereafter every three months until tumor progression.

For patients included after approval of Amendment 3 (2015-12-10), COMBIG-DC will be given as add on to standard treatment; sorafenib or Transarterial Chemoembolization (TACE).

ELIGIBILITY:
Inclusion Criteria:

* Be informed of the nature of the study and have provided written informed consent
* At least 18 years of age.
* Diagnosis of hepatocellular carcinoma according to EASL criteria or pathology.
* Radiologically measurable liver tumor(s), i.e. at least 20 mm in longest uni-dimensional diameter as measured by CT/MRI
* Not eligible for curatively aiming treatment or TACE. Tumor stage B or C according to BCLC.
* For patients included according to Amendment 3: tumour stage A, B or C according to BCLC and

  1. eligible for sorafenib treatment or having ongoing sorafenib treatment for not more than 4 weeks ant the time for inclusion or
  2. eligible for TACE or having received not more than 1 previous TACE treatment.

Exclusion Criteria:

* Performance status > ECOG 2
* Liver function according to Child-Pugh >7 points.
* Known major reaction/adverse event in connection with previously made vaccination (e.g. asthma, anaphylaxia or other serious reaction).
* Known major reaction/adverse event in connection with previous transfusions of blood products
* Active autoimmune disease requiring treatment with systemic immunosuppressive agents, e.g. inflammatory bowel disease, multiple sclerosis, sarcoidosis, psoriasis, autoimmune hemolytic anemia, rheumatoid arthritis, SLE, vasculitis, Sjögren's syndrome, scleroderma, autoimmune hepatitis, and other rheumatological diseases.
* Tested positive for HIV
* Active disease (HBV and HCV) requiring antiviral treatment
* Ongoing infection that requires treatment with antibiotics or antiviral medication
* Treatment with immunosuppressive treatments like corticosteroids (Immunosuppression (within 28 days) prior to the first injection of COMBIG-DC. Inhaled, intranasal and local steroids accepted), or mTor inhibitors within 28 days before first vaccination.
* Patients with prior history of malignancy other than HCC, within the preceding 3 years OR with relaps after complete response, except for 5 years follow-up of adequately treated in situ carcinoma without recurrences or non-melanoma skin cancer.
* Inadequate laboratory parameters, i.e.:

  1. P-Prothrombincomplex (PK) >1.4,
  2. Platelet count <50 75 x109/L
  3. Leukocyte count <3.0 x 109/L
  4. P-APT time outside normal limit
* Previous organ transplantation
* Women of Childbearing Potential (WOCBP) refusing to use adequate contraception (oral or injectable contraceptives, hormone releasing intrauterine device) throughout the study period.
* Pregnant or lactating women
* Life expectancy less than 3 months.
* Concomitant anti-tumor treatment (within 28 days) prior to the first injection of COMBIG-DC, except for sorafenib or TACE for patients included according to Amendment 3.
* For patients included according to Amendment 3: Previous systemic anti-cancer treatment.
* Investigational treatment (within 28 days) prior to the first injection of COMBIG-DC.
* Known blood dyscrasia (bleeding complication).
* Known malignancy in CNS
* Any reason that, in the opinion of the investigator, contraindicates that the patient participates in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2013-10; Primary Completion 2017-06-28 (Actual); Study Completion 2017-06-28 (Actual)

PRIMARY OUTCOMES:
Registration of adverse events as a measure of safety and tolerability | Up to 6 months after last patient's last vaccination
  * Changes in vital signs from baseline (heart rate, blood pressure, body temperature)
  * Changes in lab parameters from baseline
  * Short term worsening in ECOG and/or Child Pugh and/or MELD score
  * Local procedural injuries, assessed by MRI or ultrasound

SECONDARY OUTCOMES:
To evaluate systemic inflammatory response | Until 3 months after last vaccination
  Potential systemic release of relevant cytokines, chemokines and other inflammatory parameters in blood;IL-1R, IL-2,IL-4, IL-5, IL-6, IL-7, IL-8, IL-10, IL-12p70, IL-13, IL-17A, G-CSF. GM-CSF, IFN-gamma, MCP-1, MIP-1 beta and TNF-alpha.
To evaluate tumor control | Until 6 months after last patient's last vaccination
  * CT/MRI evaluation 3 and 6 months after first vaccination. Patients with stable disease or tumor response will continue tumor evaluation every 3rd month until progress or until last study patient has had his/her 6 month visit.
  * Measuring number of tumor specific T cells with flow cytometry after in vitro stimulation with different pools of HCC-associated tumor peptides (Alpha-feto protein (AFP), and hTERT)
  * Measuring AFP (alpha-feto protein) levels in blood
  * Measuring the level of circulating tumor cell, identified as tested positive for MICA, EpCAM, CD133, CD34, CK18
Long term changes in ECOG scores | 3 and 6 months after last vaccination
Change in body weight | 3 and 6 months after last vaccination
To evaluate systemic immunological response | Up to 3 months after last vaccination
  * Vaccine cell tracking; PBMCs will be stained with antibodies specific for one HLA class I or one HLA-class II antigen that is selectively expressed on donor vaccine cells.
  * vaccine-induced alloimmunization; screening of alloantibodies against HLA-A, B, C (MHC-class I) and HLA-DR, DQ, DP (MHC-class II) antigens
  * autoimmune events; screening of autoantibodies against autoantigens, including nuclear antigens (ANA, SSA, SSB, Sm, RNP, Scl-70, Centromeres and Jo-1) and liver parenchyma-associated autoantigens (liver-kidney microsomal antigens and mitochondrial antigens)
  * complement activation; classical/alternative complement function, C3, C4, C3d, and Factor-B.
  * immune cell occurrence and activation state; CD3+ , CD3+4+ and CD3+8+ T cells, CD19+ B-cells CD3-16+56+ NK-cells, CD3-16+56+69+ NK cells, CD3+16+56+ NKT-cells, CD3+16+56+69+ NKT-cells and CD3+HLA-DR+ T cells.
Long term changes in Quality of Life scores | 3 and 6 months after last vaccination
To evaluate immunological response | Up to 3 months after last vaccination
  * complement activation; classical/alternative complement function, C3, C4, C3d, and Factor-B.
  * immune cell occurrence and activation state; CD3+ , CD3+4+ and CD3+8+ T cells, CD19+ B-cells CD3-16+56+ NK-cells, CD3-16+56+69+ NK cells, CD3+16+56+ NKT-cells, CD3+16+56+69+ NKT-cells and CD3+HLA-DR+ T cells.
Changes in HBV, HCV virus titers | Day 8 after each injection and at the 3 and 6 months visit
  Changes in HBV, HCV virus titers vs baseline, for patients that are tested positive at screening
To study time to progress (TTP) | Measured every 3 months until progression
  TTP measured as time from first dose of COMBIG-DC until radiologically proven progress according to mRECIST.
To study overall survival (OS) | Up to 6 months after last patient's last vaccination
  OS measured as survival time from first dose of COMBIG-DC until end of study or death (whichever comes first)

OTHER OUTCOMES:
Local tissue changes in injected/non-injected tumor and surrounding tissue, assessed by MRI | 1 month after each vaccination
  An optional addition to the assessment of local procedural injuries (primary outcome).

CONTACTS AND LOCATIONS:
Overall Officials: Magnus Rizell, MD, PhD, Principal Investigator — Sahlgrenska University Hospital
Locations (1):
- Dept. of Transplantation and Liver Surgery, Sahlgrenska University Hospital, Gothenburg, Sweden

REFERENCES:
- [Derived] Rizell M, Sternby Eilard M, Andersson M, Andersson B, Karlsson-Parra A, Suenaert P. Phase 1 Trial With the Cell-Based Immune Primer Ilixadencel, Alone, and Combined With Sorafenib, in Advanced Hepatocellular Carcinoma. Front Oncol. 2019 Jan 21;9:19. doi: 10.3389/fonc.2019.00019. eCollection 2019. PMID 30719425